CLINICAL TRIAL: NCT05548556
Title: A Phase II, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Pharmacodynamics, Safety, Tolerability, Pharmacokinetics, and Efficacy of RO7204239 in Participants With Facioscapulohumeral Muscular Dystrophy
Brief Title: A Study to Evaluate RO7204239 in Participants With Facioscapulohumeral Muscular Dystrophy
Acronym: MANOEUVRE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN43703
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Facioscapulohumeral Muscular Dystrophy (FSHD)
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will complete a 4-week pre-treatment period to collect baseline movement data with a wearable device, then receive subcutaneous (SC) placebo every 4 weeks for 52 weeks. After the treatment period, participants will have the option to receive RO7204239 for an additional 52 weeks.
  Interventions: Drug: Placebo
- RO7204239 (Experimental): Participants will complete a 4-week pre-treatment period to collect baseline movement data with a wearable device, then receive SC RO7204239 every 4 weeks for 52 weeks. After the treatment period, participants will have the option to receive RO7204239 for an additional 52 weeks.
  Interventions: Drug: RO7204239

INTERVENTIONS:
Drug: Placebo — Participants will receive subcutaneous (SC) placebo every 4 weeks (Q4W)
  Arms: Placebo
Drug: RO7204239 — Participants will receive SC RO7204239 Q4W
  Arms: RO7204239

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamics, safety, tolerability, pharmacokinetics, and efficacy of RO7204239, a humanized monoclonal antibody that binds to human latent myostatin, in ambulant adult participants with facioscapulohumeral muscular dystrophy (FSHD).

ELIGIBILITY:
Inclusion Criteria:

* Genetic confirmation of FSHD1 or FSHD2
* Clinical findings consistent with FSHD
* Ability to walk unassisted
* Ricci Clinical Severity Scale score ≥ 2.5 and ≤ 4
* Agreement to maintain the same frequency and intensity of physiotherapy, occupational therapy, and other forms of exercise during the clinical study

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 17 months after the final dose of RO7204239
* Current or previous treatment (or receipt) of anti-myostatin therapies
* Treatment with any investigational therapy within 90 days prior to screening, or 5 drug-elimination half-lives of the drug, whichever is longer
* Contraindications to MRI scans
* Presence of clinically significant ECG abnormalities
* Presence of clinically significant cardiovascular disease
* Presence of clinically significant abnormal findings in echocardiography at screening, with the exception of mitral valve prolapse, which does not exclude participants from the study
* Any major illness within 1 month before screening
* Ascertained or presumptive hypersensitivity (e.g., anaphylactic reaction) to RO7204239, or to the constituents of its formulation
* History of malignancy (except in situ basal cell carcinoma of the skin and in situ carcinoma of the cervix of the uterus that have been excised and resolved with documented clean margins on pathology)
* Any clinically relevant history of anaphylactic reaction requiring inotropic support
* Any abnormal skin conditions, pigmentation, or lesions in the area intended for SC injection (abdomen) and that would prevent visualization of potential injection-site reactions to RO7204239
* Immobilization, surgical procedures, fracture, or trauma to the upper or lower limbs within 90 days prior to screening or longer, if judged by the investigator that it may affect motor function assessment
* Any planned surgery that may affect a participant's motor function assessment, including participants who have had surgery of scapular fixation within the 12 months preceding screening or that are planned during the study
* Use of the following medications within 90 days prior to enrollment: salbutamol or another β2-adrenergic agonist taken orally; creatine; recombinant human growth hormone; recombinant human insulin growth factor-1; testosterone, oxandrolone, or other anabolic steroid; chronic oral or parenteral use of corticosteroids (inhaled corticosteroid use is allowed) unless required to manage injection reactions;agents anticipated to increase or decrease muscle volume or strength

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in contractile muscle volume (CMV) of quadriceps femoris muscles as assessed by magnetic resonance imaging (MRI) bilaterally | Week 52
Percentage of participants with adverse events (AEs) | Up to 2.5 years

SECONDARY OUTCOMES:
Change from baseline in serum concentration of total latent myostatin | Through 2 years
Change from baseline in serum concentration of free latent myostatin | Through 2 years
Change from baseline in serum concentration of mature myostatin | Through 2 years
Percent change from baseline in CMV of 36 muscles based on whole body MRI | Weeks 28 and 52
Change from baseline in fat fraction of 36 muscles based on whole body MRI | Weeks 28 and 52
Percent change from baseline in CMV of quadriceps femoris muscles as assessed by MRI bilaterally | Week 28
Change from baseline in fat fraction of quadriceps femoris muscles as assessed by MRI bilaterally | Weeks 28 and 52
Percent change from baseline in CMV of tibialis anterior muscles as assessed by MRI bilaterally | Weeks 28 and 52
Change from baseline in fat fraction of tibialis anterior muscles as assessed by MRI bilaterally | Weeks 28 and 52
Percent change from baseline in CMV of biceps brachii muscles as assessed by MRI bilaterally | Weeks 28 and 52
Change from baseline in fat fraction of biceps brachii muscles as assessed by MRI bilaterally | Weeks 28 and 52
Percent change from baseline in contractile cross-sectional area (CSA) of skeletal muscle in the proximal lower limb muscles as assessed by MRI bilaterally | Weeks 28 and 52
Change from baseline in fat fraction of proximal lower limb muscles as assessed at a single mid-femur slice bilaterally by MRI | Weeks 28 and 52
Serum concentration of RO7204239 | Through 2 years
Maximum serum concentration (Cmax) of RO7204239 | Through 2 years
Area under the concentration-time curve (AUC) of RO7204239 | Through 2 years
Trough concentration (Ctrough) of RO7204239 | Through 2 years
Percentage of participants with anti-drug antibodies (ADAs) | Baseline up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United States (5):
  - University of Irvine Medical Center (UCIMC), Orange, California
  - Regents of the University of Colorado, Aurora, Colorado
  - University of Kansas Medical Center, Fairway, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- Rigshospitalet, København Ø, Denmark
- Italy (2):
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Asst Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
- United Kingdom (2):
  - National Hospital for Neurology and Neurosurgery,, London
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing